CLINICAL TRIAL: NCT03727295
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of Idebenone in the Treatment of Early-stage Parkinson's Disease With Motor and Non-motor Symptoms
Brief Title: Idebenone Treatment of Early Parkinson's Diseasesymptoms
Acronym: ITEP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZDX-1
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-05

CONDITIONS: Oxidative Stress is an Important Cause of Parkinson's Disease
MeSH Terms: interventions — idebenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The control group 1 (Experimental): 60 cases, idebenone 180mg/d, 3 times / day, oral
  Interventions: Drug: Idebenone/placebo
- The control group 2 (Experimental): 60 cases, idebenone 360mg/d, 3 times / day, oral
  Interventions: Drug: Idebenone/placebo
- The placebo group (Placebo Comparator): 60 cases, placebo, 3 times / day, oral
  Interventions: Drug: Idebenone/placebo

INTERVENTIONS:
Drug: Idebenone/placebo — The two control group will be given Idebenone in two different doses，and the placebo group will be given placebo

SUMMARY:
On May 30,2018 ,Investigators intend to conduct a multicenter, randomized, double-blind, placebo-controlled study of idebenone in the treatment of early-stage Parkinson's disease with motor and non-motor symptoms which is to observe the therapeutic effect of idebenone on motor symptoms and non-motor symptoms in patients with early Parkinson's disease。

DETAILED DESCRIPTION:
This clinical trail was a multicenter, parallel, randomized, double-blind, placebo-controlled study led by Professor Liu Chunfeng from the Second Affiliated Hospital of Suzhou University which consisted of 15 sub-centers with a total of 180 subjects.

This clinical study is divided into two phases:

The first stage: double-blind period, 24 weeks. Three queues containing idebenone 180 mg/d,360 mg/d and placebo.

The second stage: open label extension period, 24 weeks. All enrolled participants continued to take idebenone 180 mg/d to study the long-term effects of idebenone.

ELIGIBILITY:
Inclusion Criteria:

* (1) Male or female, age > 30 years old, ≤ 80 years old;
* (2) Conforms to the "Diagnostic Criteria for Parkinson's Disease" developed by the 2015 International Association of Sports Disabilities (MDS);
* (3) Patients with early Parkinson's disease, duration <3 years, Hoehn-Yahr classification:1-3, MMSE scale score ≥ 24 points;
* (4)Receiving a stable dose of dopamine agonist or monoamine oxidase type B inhibitor for treatment before the enrollment;
* (5) The subjects need to sign the Informed Consent Form（ICF）

Exclusion Criteria:

* (1)Patients with disturbance of consciousness, aphasia and mental illness; patients with major depression (HAD scale score ≥ 15 points)
* (2)Patients with Parkinson's superimposition syndrome and patients with secondary Parkinson's syndrome (hepatolenticular degeneration, hepatic encephalopathy, cerebellar disease, hydrocephalus, parathyroid disease, etc.)
* (3)Patients who have long-term use of dopamine blockers (such as potent neuroleptics, sibutramine, reserpine, metoclopramide, etc.);
* (4)Patients who have taken coenzyme Q10 or idebenone within three months;
* (5) Patients taking amantadine and levodopa need to stop taking the drug for more than one month before the enrollment;
* (6)Patients with severe cardiopulmonary dysfunction, liver and kidney dysfunction (more than 3 times normal);
* (7)Patients who cannot cooperate with the neuropsychological test;
* (8) Patients with poor compliance, not following the prescribed treatment regimen.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy on motor symptoms and non-motor symptoms | 48weeks
  UPDRS-III Hoehn-Yahr classification Olfactory function test Anxiety and depression: Anxiety and Depression Scale (HAD)

IPD SHARING:
Plan to Share IPD: Undecided